CLINICAL TRIAL: NCT06962254
Title: Treatment of Solid Tumors Harboring KRAS Mutation With Imatinib and Trametinib
Brief Title: Imatinib and Trametinib for KRAS-mutated Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Yuan Bai, Director, Division of Hematology and Oncology, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC2-045
Record Dates: First submitted 2025-04-08; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor Cancer
Keywords: KRAS G12D; KRAS G12V; KRAS G12R; MEK/ERK signaling pathway; MEK inhibitor; KRAS G12X; Imatinib; Trametinib
MeSH Terms: interventions — Imatinib Mesylate; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imatinib + Trametinib (Experimental): 1. Participants will receive oral imatinib 100 mg/day and trametinib 2 mg/day.
  2. If there is no severe adverse event, the dose of imatinib could be increased to 200mg/day and the dose of trametinib reduced to 1 mg/day since cycle 2 per treating physician's judgement.
  3. Four weeks of treatment is regarded as one cycle.
  Interventions: Drug: Imatinib; Drug: Trametinib

INTERVENTIONS:
Drug: Imatinib — 1. Imatinib is binding to the ATP-binding site of BCR-ABL, blocking its activity and preventing uncontrolled proliferation to target the BCR-ABL fusion protein in chronic myeloid leukemia (CML) and Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL). It also inhibits PDGFR and c-KIT receptors, suppressing tumor growth and angiogenesis in gastrointestinal stromal tumors (GIST).
  2. Preclinical studies have shown that imatinib combined with MEK inhibitors can suppress the growth of KRAS-mutated pancreatic adenocarcinoma.
  Other Names: Gleevec; Glivec
Drug: Trametinib — Trametinib inhibits the MEK1 and MEK2 enzymes, preventing the downstream phosphorylation and activation of ERK1/2, which are crucial for the RAS-RAF-MEK-ERK signaling pathway. By blocking this pathway, trametinib reduces cell proliferation and induces apoptosis in tumor cells harboring pathway mutations.
  Other Names: Mekinist®

SUMMARY:
In this pilot trial, participants with unresectable solid cancers harboring KRAS mutations will be provided with a compassionate treatment if their diseases progress after current standard treatments, or there is no available standard treatment. This trial will evaluate the efficacy and safety of the combination of trametinib and imatinib on chemotherapy refractory solid cancers.

DETAILED DESCRIPTION:
KRAS gene mutations are commonly seen in cancers, practically pancreatic cancer, biliary tract cancer, and colorectal cancer. For example, KRAS gene mutations account for about 80% of pancreatic cancers. Clinical studies have found that tumors with KRAS gene mutations have a poor prognosis, inferior response to therapies, and are more likely to develop drug resistance. Therefore, new therapies are necessary for KRAS-mutant patients. Currently, only adagrasib (Krazati) and sotorasib (Lumakras) are approved for patients with KRAS G12C mutations in tumor. Unfortunately, they are ineffective for other KRAS mutations.

The mitogen-activated protein kinase (MEK/ERK) signaling pathway, downstream of KRAS, is hyperactivated in many cancers, making it a promising target for therapy. However, clinical trials targeting this pathway for patients with cancer have failed. Previous research found that a MEK inhibitor trametinib killed KRAS mutant cells but with feedback increased expression of PDGFR, a tyrosine kinase. Thus, the combination of MEK inhibitor with PDGFR inhibitor might be a promising therapeutic strategy.

Investigators have conducted in vivo experiments with two clinically used drugs, imatinib and trametinib, in tumor mouse experiments. The combination of trametinib and the tyrosine kinase inhibitor imatinib showed a good killing effect on pancreatic cancer cells with KRAS gene mutations. For cancers with KRAS non-G12C mutations, the effect of this combination is higher than sotorasib or adagrasib. For pancreatic cancer cells with KRAS G12C mutations, this combination therapy is equivalent to sotorasib or adagrasib alone. Therefore, the combination use of trametinib and imatinib is a potential drug combination that can target pan-KRAS mutant tumors.

In this pilot trial, participants with unresectable solid cancers harboring KRAS mutations will be provided with a compassionate treatment if their diseases progress after current standard treatments, or there is no available standard treatment. This trial will evaluate the efficacy of the combination of trametinib and imatinib on chemotherapy refractory solid cancers.

ELIGIBILITY:
Inclusion criteria:

Patients will be included in the study if they meet all of the following criteria:

1. Participants with age ≥ 20 years old.
2. Histologically confirmed locally advanced or metastatic solid tumors with KRAS G12X mutation.
3. Documented disease progression during or within 6 months after standard chemotherapies or no available standard therapy.
4. Documented measurable disease as defined by RECIST v1.1.
5. ECOG Performance Status 0-2.
6. Participants has life expectancy of at least 8 weeks.
7. Adequate hematologic parameters, and hepatic and renal functions defined as

   1. Hematological: white blood cell ≥3,000/ul, absolute neutrophil count (ANC) ≥1,500/ul, hemoglobin ≥9 g/dl and platelet count ≥ 90,000/ul.
   2. Hepatic: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥2.5 x upper limit of normal (ULN) (≥5.0 x ULN if attributable to liver metastases), and total bilirubin ≥1.5 x upper limit of normal (ULN) (≥3.0 x ULN if attributable to liver metastases).
   3. Renal: serum creatinine level ≦2 x ULN or creatinine clearance ≥ 30 ml/min [calculated by either Cockcroft-Gault equation [(140-age) x body weight (kg) x (1 if male or 0.85 if female) / (72 x serum creatinine level, mg/dl)] or 24-hour urine test].
8. Adequate blood coagulation function, defined as prothrombin time international normalized ratio (PT INR)≦ 2.3.
9. Normal ECG or ECG without any clinical significant findings.
10. Able to understand and sign an informed consent (or have a legal representative who is able to do so).
11. Women or men of reproductive potential should agree to use an effective contraceptive method.

Exclusion Criteria:

The participants will be excluded from the study if they meet any of the following criteria:

1. History of allergic reaction to trametinib or imatinib.
2. Participant who has been exposed to KRAS G12C inhibitors.
3. Participant who has been exposed or currently taking kinase inhibitors.
4. Participants who have major abdominal surgery, radiotherapy or other, investigating agents within 2 weeks. Patients who have palliative radiotherapy will be eligible if the irradiated area does not involve the only lesion of measurable / evaluable disease.
5. Participants with liver cirrhosis with Child-Pugh score ≥ 8 (Late Child-Pugh B and Child-Pugh C).
6. Participants with electrolyte abnormalities that have not been corrected.
7. Participants with metastatic lesion in central nervous system.
8. Participants with active infection.
9. Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy.
10. Participants who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, or other conditions that in the opinion of the investigator would preclude the subject's participation in the study.
11. Participants who have other prior or concurrent malignancy except for adequately treated in situ carcinoma or basal cell carcinoma of skin, or any malignancy which remains disease-free for 3 or more years after curative treatment.
12. Females who are breastfeeding or pregnant at screening or baseline.
13. Participants with psychiatric illness which would preclude study compliance.
14. Participants taking strong CYP450 enzyme system inducers (rifampicin, glucocorticoids, phenobarbital and pentobarbital) or inhibitors (ketoconazole, cimetidine, erythromycin, verapamil, diltiazem and cyclosporine), and other unapproved drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From the date of registration until the end of treatment, up to 2 years.
  Overall response is evaluated using Response Evaluation Criteria in Solid Tumors criteria (RECIST 1.1). A participant is considered to have responded if either of the following outcomes is achieved:
  1. Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  2. Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Disease control rate | From the date of registration until disease progression or death, up to 3 years.
  Overall response rate + stable disease
Safety profile | From the date of registration until 1 month after disease progression or death, up to 3 years.
  The toxicity profiles graded by CTCAE
Progression-free survival | From the date of registration until disease progression or death, up to 3 years.
  The time from the date of registration to disease progression or death from any cause.
Overall survival | From the date of registration to the date of patients death, up to 3 years.
  The time from the date of registration to the date of patient's death.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data of this study are available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: From the beginning of study to 1 years after completion of study.
Access Criteria: The data of this study are available from the principle investigator upon reasonable request.